CLINICAL TRIAL: NCT07365943
Title: The Effect of Forgiveness-based Motivational Interviewing on Death Anxiety, Life Satisfaction, and Forgiveness Disposition in Patients With COPD: A Randomized Controlled Trial
Brief Title: The Effect of Forgiveness-based Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer USLU (Other)
Responsible Party: Sponsor-Investigator, Ömer USLU, Dr. Ömer USLU, PhD-Principal Investigator, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERVE-RCT-2025-COPD
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Nursing; Psychoeducation; COPD (Chronic Obstructive Pulmonary Disease); Forgiveness
Keywords: Death anxiety; forgiveness; life satisfaction; COPD; motivational interviewing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Necrophobia; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study used a pretest-posttest-follow-up randomised controlled experimental method. Participants were randomly assigned to either the experimental group (forgiveness based motivational interviewing) or the control group with no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- forgiveness-based motivational interviewing (Experimental): Participants will receive an 6-session forgiveness-based motivational interviewing
  Interventions: Other: forgiveness-based motivational interviewing; Other: Control
- Control (No Intervention): Throughout the study, the forgiveness-based motivational interviewing was applied only to the experimental group, and no intervention was performed in the control group

INTERVENTIONS:
Other: forgiveness-based motivational interviewing — The forgiveness-based motivational interviewing was administered face-to-face, with each session lasting 40-60 minutes, scheduled twice a week over a three-week period (a total of six sessions).
  Arms: forgiveness-based motivational interviewing
Other: Control — no intervention was performed in the control group
  Arms: forgiveness-based motivational interviewing

SUMMARY:
This study aimed to examine the effect of forgiveness-based motivational interviewing on death anxiety, life satisfaction, and forgiveness disposition in patients with COPD. A randomized controlled experimental design with pretest, posttest, and one-month follow-up measurements was employed. The study sample consisted of 30 patients (experimental group: 15; control group: 15). The experimental group received forgiveness-based motivational interviewing, whereas no intervention was provided to the control group. Data were collected using a personal information form, the Death Anxiety Scale, the Life Satisfaction Scale, and the Forgiveness Scale. The findings revealed that, in the posttest and follow-up measurements, the experimental group had significantly lower mean scores on the Death Anxiety Scale compared to the control group (p<0.05). Furthermore, the experimental group demonstrated significantly higher mean scores on the Life Satisfaction Scale and the Forgiveness Scale in the posttest and follow-up measurements than the control group (p<0.05). This study concluded that forgiveness-based motivational interviewing effectively reduces death anxiety while enhancing life satisfaction and forgiveness disposition in patients with COPD. Therefore, implementing motivational interviewing for patients is recommended.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a global chronic respiratory disease that arises from a combination of genetic and environmental factors, predominantly due to smoking and air pollution.As the disease progresses, symptoms such as dyspnoea, cough, and sputum production emerge, leading to several complications, including fatigue, insomnia, social withdrawal, and anxiety. The persistent presence of these symptoms can result in intense death anxiety among COPD patients. Studies on COPD patients in the literature suggest that the prolonged duration of the disease, continuous medication use, and the burden of disease-related symptoms negatively impact their quality of life, ultimately reducing their life satisfaction. This decline in life satisfaction can, in turn, give rise to a diminished sense of hope for the future and an escalation in death anxiety. Moreover, COPD patients frequently encounter emotional distress during treatment and care, undergo a critical reassessment of their past lives, and grapple with feelings of guilt and regret. The management of these emotions can be arduous. In this context, the concept of forgiveness emerges as a potential mitigating factor for the adverse emotional effects of the disease. Forgiveness is not about denying the pain and consequences of a distressing experience but rather an effort to replace feelings of anger, resentment, and bitterness with compassion, empathy, and kindness. To date, no studies have specifically examined forgiveness training for COPD patients; however, previous research indicates that motivational interviewing has positive effects on various patient populations. Motivation can be defined as an internal state influenced by external factors. Motivational interviewing is a client-centred and encouraging approach that helps individuals explore and resolve ambivalence to facilitate behaviour change. Motivational interviewing not only supports behavioural and lifestyle changes in patients but also enhances their adherence to treatment. Beyond the necessity of treating physical symptoms in individuals with chronic diseases like COPD, the need for psychological support underscores the importance of consultation-liaison psychiatry. Consultation-liaison psychiatry (CLP) nurses do not merely provide care services; they also assume advisory and educational roles by conducting individual or group psychoeducation sessions. CLP nurses should support patients in expressing emotions such as anger, guilt, sadness, and regret, strengthen their coping mechanisms, mobilise effective support systems, and increase awareness of the impact of these emotions on their lives. In consideration of the role of CLP nurses, it can be posited that forgiveness-based motivational interviewing for COPD patients may prove efficacious in reducing death anxiety, increasing life satisfaction, and enhancing forgiveness tendencies, while concomitantly addressing their need for care, education, and counselling.

ELIGIBILITY:
Inclusion Criteria:

* They must be 18 years of age or older,
* Possess sufficient mental capacity and communication skills to follow the study guidelines, be literate,
* Have a diagnosis of COPD,
* Have been hospitalized in the pulmonary diseases unit between June and September 2024.

Exclusion Criteria:

* Determined having communication barriers due to disease symptoms,
* Experiencing dyspnea at a level that prevents cooperation
* Having a chronic psychiatric disorder that would interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Death Anxiety Scale | Baseline (pretest), 3 weeks (posttest) and one month after the posttest
  The scale is a unidimensional, dichotomous Likert-type instrument consisting of 15 items that assess an individual's anxiety related to their own death and the risk of dying. Each item is answered as "yes" or "no," where a "yes" response for the first nine items and a "no" response for the remaining six items receive one point. The total score ranges from 0 to 15, with higher scores indicating greater death anxiety.

SECONDARY OUTCOMES:
Forgiveness scale | Baseline (pretest), 3 weeks (posttest) and one month after the posttest
  Forgiveness Scale, developed by Ersanlı and Batık, designed to measure individuals' levels of self-forgiveness and forgiveness of others. The scale is scored from "strongly disagree" to "strongly agree," with higher scores indicating higher levels of forgiveness.

OTHER OUTCOMES:
Life satisfaction scale | Baseline (pretest), 3 weeks (posttest) and one month after the posttest
  The scale consists of a single dimension with five items, rated on a five-point Likert scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). The total score ranges from 5 to 25, with higher scores indicating higher life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Şahin, PhD, RN, Principal Investigator — Bergama Necla Mithat Öztüre State Hospital
Locations (1):
- Bergama Necla Mithat Öztüre State Hospital, Izmir, Bergama, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to ethical and institutional restrictions. The dataset includes sensitive health information from postpartum women, and the informed consent process did not include permission for public data sharing. Therefore, in accordance with privacy regulations and ethical committee requirements, IPD will not be made available to other researchers

REFERENCES:
- See also: Bergama Necla Mithat Öztüre State Hospital — https://bergamadh.saglik.gov.tr